CLINICAL TRIAL: NCT05061121
Title: Effect of Sustained Natural Apophyseal Glides and Myofascial Release on Chronic Non-specific Neck Pain : Randomized Controlled Trial
Brief Title: Effect of Sustained Natural Apophseal Glides and Myofascial Release on Chronic Non-specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amal Ahmed Mohamed Morsi Abdel-Baky, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNAGs and MFR
Record Dates: First submitted 2021-08-31; First posted 2021-09-29 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Neck Pain
Keywords: CNSNP; SNAGs; MFR
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Design of the study:
  Single-blinded randomized controlled trial design. Patients will be randomly assigned into 3 equal groups using the statistical package for social science (SPSS 20).
  Group A (Mulligan's SNAGs) Group B (Myofascial release) Group C (Mulligan's SNAGs + Myofascial release)
Who Masked: Participant
Masking Description: assigned randomly into Three equal groups the by using permuted block method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sustained natural apophyseal glides (Experimental): Investigate the short- and mid-term effects of Mulligan's SNAGs on pain intensity, pain pressure sensitivity, cervical function, range of motion (ROM) and postural stability in CNSNP patients
  Interventions: Other: combined effect
- Myofascial release (Experimental): Investigate the short- and mid-term effects of Myofascial release on pain intensity, pain pressure sensitivity, cervical function, range of motion (ROM) and postural stability in CNSNP patients
  Interventions: Other: combined effect
- sustained natural apophyseal glides in addition to myofascial release (Experimental): Investigate the short- and mid-term effects of Mulligan's SNAGs combined with Myofascial release on pain intensity, pain pressure sensitivity, cervical function, range of motion (ROM) and postural stability in CNSNP patients
  Interventions: Other: combined effect

INTERVENTIONS:
Other: combined effect — Compare the short- and mid-term effects of Mulligan's SNAGs, Myofascial release, and their combination on pain intensity, pain pressure sensitivity, cervical function, range of motion (ROM) and postural stability in CNSNP patients

SUMMARY:
The aim of investigator's study is to combine and compare the two scientifically approved therapies for the CNSNP to investigate the short term and mid-term changes of the combination of these two manual techniques concerning pain, function, range of motion ROM and postural stability.

DETAILED DESCRIPTION:
Neck pain NP is a recognized medical and socioeconomic problem, which is responsible for high treatment costs, sick leave, and individual suffering, in addition to being one of the main reasons for people to seek health care services .NP is widely spread in healthcare centers with a prevalence estimation of 288.7 million, in North Africa and the Middle East ranged between 3917.7 to 5022.4 per 100 000 populations in 2017. NP with symptoms duration exceeding 12 weeks is considered chronic.

Individuals who have chronic non-specific neck pain CNSNP have less quality of life, and more pain interference in their life. More over studies showed that patients with CNSNP subjects have poorer postural control than healthy subjects.

Alteration of the proprioception of the neck muscles and joints that play a master role in the cervical joint position and motor control of the head could be the primary cause of CNSNP . Studies have evaluated the effect of different manual techniques in cases of CNSNP checking mainly usefulness and effectiveness of these interventions on this clinical condition. However, there is less evidence in literature investigating the short and mid-term changes of these techniques.

Manual therapy, is a physical treatment primarily used by physical therapists, occupational therapists, manipulative therapy to treat musculoskeletal pain and disability; it is most commonly includes kneading , manipulation of the muscles and mobilization of joints .Many Studies investigating the effectiveness of manual therapies on CNSNP ,proving reduction of spinal excitability and pain sensitivity, enhancement of function and range of motion.

Brian Mulligan techniques are widely used for joint dysfunction by growing number of therapists and are an important addition to the field of Manual Therapy. Literature reveals many and diverse treatment approaches for chronic neck pain. Sustained natural apophyseal glides SNAGs are pain free spinal manual therapy treatment techniques involving concurrent accessory joint gliding and active physiological movement, with overpressure at end range, which are utilized for painful movement restrictions of the spine.

Mulligan's SNAGs is one of the most statistically proved in many studies that manual therapy technique affects proprioception, function, range of motion, pain.

On the other hand, Myofascial release which is a form of soft tissue therapy that is intended to reduce pain and increase mobility in patients that are suffering from chronic pain conditions. Myofascial release has shown effectiveness in reducing mechanical neck pain and in improving functional abilities by freeing restrictions of movement that originate in the soft tissues of the body.

Furthermore, as the focus of most previous studies has been to examine compare mulligan's SNAGs and Myofascial release separately, studies on their combination effects have been largely ignored. Both two techniques have shown efficacy, but since SNAGS and Myofascial release are different mechanisms of action, the time of their effects and their progression could be different.

The aim of investigators' study is to combine and compare the two scientifically approved therapies for the CNSNP to investigate the short term and mid-term changes of the combination of these two manual techniques concerning pain, function, range of motion ROM and postural stability.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 20-45 years
* Current neck pain
* Neck pain continued for at least the last 12 week
* Pain with no obvious organic or pathologic cause.
* The patients diagnosed as chronic non-specific neck pain through an orthopedic specialist, diagnostic investigations including X rays and MRI failed to show obvious pathological findings

Exclusion Criteria:

* Irradiated neck pain
* Neck pain associated with vertigo
* Osteoporosis
* Diagnosed psychological disorders
* Vertebral fractures
* Tumors
* Diagnosed metabolic diseases
* Previous neck surgery
* Red flags (night pain, severe muscle spasm, loss of
* involuntary weight, symptom mismatch)
* Physiotherapeutic treatment continued in the last 3 months

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
pain intensity VAS | 15 mins
  visual analogue scale ,The pain VAS is a continuous scale formed of a horizontal (HVAS) or vertical (VVAS) line, 100 mm in length, ended with 2 verbal pain descriptor on either end one for each symptom extreme; "no pain" at the most left side of the line (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 /100-mm scale) on the rightest end
Pressure pain threshold PPT | 30 mins
  pressure algometer ,The PPT represents a hybrid test, falling somewhere between self-reported paper-and-pencil type tools and objective diagnostic techniques
function | 15 mins
  Neck Disability Index (NDI) This index consists of ten sections, including seven sections related to activities of daily living, two sections related to pain, and one section related to concentration. The score for each section is from 0 to 5, with 0 representing the highest level of function and 5 representing the lowest level of function. Total NDI-TH scores are shown as a percentage. A high score corresponds to a higher degree of disability. The internal consistency of the NDI-TH is high.
Range of motion | 30 mins
  Cervical range of motion device (CROM) The CROM device is a reliable outcome tool for measuring upper cervical rotation. The clinical implications of these findings suggest that therapists can utilize the CROM device to more completely examine all planes of upper and full cervical mobility. It may also assist in identifying upper cervical ROM limitations associated with underlying cervical pathology or motion dysfunction
postural stability | 30 mins
  Biodex Balance System (BBS) The Biodex balance system (BBS) uses a circular platform that is free to move in the anterior-posterior and medial-lateral axes simultaneously, which permits three measures to be obtained: an overall stability index (OSI), an anterior-posterior stability index (APSI), and a medial-lateral stability index (MLSI) will measure OSI ,APSI ,and MLSI

CONTACTS AND LOCATIONS:
Locations (1):
- Misr University For Science and Technology, El-Sheikh Zayed City, Giza Governorate, Egypt

REFERENCES:
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399
- [Background] Binder A. The diagnosis and treatment of nonspecific neck pain and whiplash. Eura Medicophys. 2007 Mar;43(1):79-89. PMID 17369782
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164
- [Background] Gonzalez Rueda V, Lopez de Celis C, Barra Lopez ME, Carrasco Uribarren A, Castillo Tomas S, Hidalgo Garcia C. Effectiveness of a specific manual approach to the suboccipital region in patients with chronic mechanical neck pain and rotation deficit in the upper cervical spine: study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2017 Sep 5;18(1):384. doi: 10.1186/s12891-017-1744-5. PMID 28870191